CLINICAL TRIAL: NCT05651971
Title: A Prospective, Observational Study of the Anatomical Localization of the Inferior Mesenteric Artery in Relation to the Left Colonic Artery During Laparoscopic Radical Surgery for Rectal Cancer
Brief Title: The Anatomical Localization of the Inferior Mesenteric Artery in Relation to the Left Colonic Artery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202201-18
Record Dates: First submitted 2022-11-16; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: measurement group — Measurement of the distance between the origin of LCA (left colonic artery，LCA) and IMA (inferior mesenteric artery，IMA) root and the distance between IMA and IMV (inferior mesenteric vein，IMV) at the origin of LCA in rectal cancer patients

SUMMARY:
1. To observe and measure the distance between the origin of LCA (left colonic artery，LCA) and IMA (inferior mesenteric artery，IMA) root and the distance between IMA and IMV (inferior mesenteric vein，IMV) at the origin of LCA in rectal cancer patients. Statistical analysis of intraoperative measured data, on the basis of the original anatomical relationship, to achieve anatomical localization of quantitative and accurate, for the preservation of LCA laparoscopic radical resection of rectal cancer to provide a strong anatomical basis.
2. The operation time, 253 lymph node dissection time, intraoperative blood loss, postoperative anal exhaust time, postoperative feeding time, postoperative hospital stay, postoperative ischemic colitis rate and postoperative anastomotic leakage rate of patients with laparoscopic radical resection of rectal cancer with preservation of LCA were recorded. The surgical efficacy and clinical significance of laparoscopic radical resection of rectal cancer with preservation of LCA were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of rectal cancer (T2-4a, N- / +, M0) ; Laparoscopic radical resection of rectal cancer and preservation of LCA Patients and their families agree to participate in the clinical study

Exclusion Criteria:

* Those who had a history of lower abdominal surgery and could not undergo laparoscopic surgery LCA vascular absence was found during operation combined with other malignant tumors pregnant or lactating patients Combined with severe mental illness Severe diseases of the blood system, coagulation dysfunction ; Preoperative assessment of heart, lung and brain function, unable to tolerate surgery.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The age was between 18 and 75 years old, and the pathological diagnosis was rectal cancer (T2-4a, N- / +, M0)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Distance between LCA and IMA | intraoperative
  Measurement of the distance between the origin of LCA (left colonic artery，LCA) and IMA (inferior mesenteric artery，IMA) root
The distance from LCA to IMA and IMV | intraoperative
  Measurement of the distance between IMA and IMV (inferior mesenteric vein，IMV) at the origin of LCA

SECONDARY OUTCOMES:
operation time | intraoperative
  From the beginning of anesthesia to the patient leaving the operating room
253 lymph node dissection time | intraoperative
  Record the time required to dissection 253 lymph node
intraoperative blood loss | intraoperative
  Record intraoperative bleeding
exhaust time | Within one week after operation
  Record the time of patient's first exhausting time after operation
postoperative feeding time | Within one week after operation
  Record the time of the patient's first meal after operation
postoperative hospital time | Within two weeks after operation
  Record the days from surgery to discharge
postoperative anastomotic leakage rate | One month after operation
  Record the situation of patient's anastomotic leakage

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Gastriontestinal Department, Tang-Du of Fourth Medical University, Xi’an, Shanxi, China